CLINICAL TRIAL: NCT01695720
Title: Trial Comparing VisionScope Imaging (VSI) With Magnetic Resonance Imaging (MRI) in the Diagnosis of Suggestive Clinical Symptoms for Meniscus and Articular Cartilage Injuries in the Knee
Brief Title: Clinical Efficacy Study Comparing VisionScope Imaging (VSI) to Magnetic Resonance Imaging (MRI) in Injuries of the Knee
Acronym: VSI-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VisionScope Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VisionScope VSI-001
Record Dates: First submitted 2012-09-13; First posted 2012-09-28 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Meniscus Tears; Loose Bodies; Articular Osteoarthritis; Articular or Capsular Trauma
Keywords: Knee Injuries; Meniscus Injuries; Articular Cartilage Injuries; Orthopaedic Diagnostic; Magnetic Resonance Imaging
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VisionScope Imaging (VSI) Exam (Experimental): A VisionScope Imaging (VSI) Exam is diagnostic arthroscopic procedure. Through a natural or surgical opening, an endoscope is inserted through a cannula to illuminate and visualize the interior cavity of a joint.
  Interventions: Procedure: VisionScope Imaging (VSI) Exam

INTERVENTIONS:
Procedure: VisionScope Imaging (VSI) Exam — The VisionScope Imaging (VSI) Exam [the system itself] is indicated for use in diagnostic and operative arthroscopic and endoscopic procedures to provide illumination, visualization, and the capture of still and motion pictures of an interior cavity of the body through a natural or surgical opening.

SUMMARY:
The purpose of the study is to accumulate efficacy data on VisionScope Imaging (VSI) for pre-operative diagnosis of certain knee injuries (meniscal and articular cartilage injuries). The study will compare VSI's accuracy to MRI's in diagnosing the same injuries.

The hypothesis is the VisionScope Imaging system will be able to provide direct visualization and diagnostic images of inside the joint capsule space without fluid distention in the knee. This study will provide valuable feedback on the ability of the VisionScope system to provide physicians with the information they need to make a definitive diagnosis.

DETAILED DESCRIPTION:
The primary objective of this study is to accumulate efficacy data on the VisionScope Imaging System (VSI) for pre-operative diagnoses when it is used to provide illumination and visualization of articular cavities. The study will analyze the VisionScope system's accuracy compared to MRI in diagnosing and confirming meniscus tears, chondral defects, loose bodies, minor arthritis, and/or any articular or capsular trauma.

The hypothesis of the study is that the VisionScope System will be able to obtain direct visualization and diagnostic images of the intercapsular space without fluid distention in the knee. This study will provide feedback on the ability of the VisionScope system to potentially eliminate the need for MRI scans. Additionally, a cost-analysis comparison between the use of VSI vs. MRI for the diagnosis of orthopaedic knee injuries will be conducted. Finally, the study will help develop an algorithm of potential use for the VSI system in the management of knee pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Suspected meniscal injuries to the knee
* Suspected articular cartilage injuries to the knee

Exclusion Criteria:

* Acute traumatic hemarthroses and/or concomitant ligament injury
* Active systemic infection
* Allergy to silicone or any medication used during the procedure
* Enrollment in another pharmacological or medical device study
* Institutionalized persons, prisoners and persons with decisional incapacity
* Investigator's own students and employees

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy | 1 day
  Diagnostic accuracy will be assessed during the time of the procedure. There will be no patient followup in this study. Radiologists, post procedure, will compare/contrast the diagnostic findings of a patient's MRI, VSI and Dx Arthroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Gill, IV, MD, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (7):
  - Kerlan-Jobe Orthopaedic Foundation, Los Angeles, California
  - Stanford School of Medicine, Redwood City, California
  - Santa Monica Orthopaedic & Sports Medicine Group (SMOG), Santa Monica, California
  - Andrews Research and Education Institute, Gulf Breeze, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Texas SouthWestern, Dallas, Texas
  - Mansfield Orthopaedics (Copley Hospital), Morrisville, Vermont

REFERENCES:
- [Background] Rheumatology 2000; 39: 700-706, British Society for Rheumatology
- [Background] Ryzewicz M, Peterson B, Siparsky PN, Bartz RL. The diagnosis of meniscus tears: the role of MRI and clinical examination. Clin Orthop Relat Res. 2007 Feb;455:123-33. doi: 10.1097/BLO.0b013e31802fb9f3. PMID 17279041
- [Background] Ruwe PA, McCarthy SM. Cost effectiveness of magnetic resonance imaging of the knee. Magn Reson Imaging Clin N Am. 1994 Aug;2(3):475-9. PMID 7489301
- [Background] Rappeport ED, Wieslander SB, Stephensen S, Lausten GS, Thomsen HS. MRI preferable to diagnostic arthroscopy in knee joint injuries. A double-blind comparison of 47 patients. Acta Orthop Scand. 1997 Jun;68(3):277-81. doi: 10.3109/17453679708996701. PMID 9246993
- [Background] Rangger C, Klestil T, Kathrein A, Inderster A, Hamid L. Influence of magnetic resonance imaging on indications for arthroscopy of the knee. Clin Orthop Relat Res. 1996 Sep;(330):133-42. doi: 10.1097/00003086-199609000-00016. PMID 8804283
- [Background] De Smet AA, Mukherjee R. Clinical, MRI, and arthroscopic findings associated with failure to diagnose a lateral meniscal tear on knee MRI. AJR Am J Roentgenol. 2008 Jan;190(1):22-6. doi: 10.2214/AJR.07.2611. PMID 18094289
- [Background] Halinen J, Koivikko M, Lindahl J, Hirvensalo E. The efficacy of magnetic resonance imaging in acute multi-ligament injuries. Int Orthop. 2009 Dec;33(6):1733-8. doi: 10.1007/s00264-008-0689-6. Epub 2008 Dec 3. PMID 19050885
- [Background] Mandelbaum BR, Finerman GA, Reicher MA, Hartzman S, Bassett LW, Gold RH, Rauschning W, Dorey F. Magnetic resonance imaging as a tool for evaluation of traumatic knee injuries. Anatomical and pathoanatomical correlations. Am J Sports Med. 1986 Sep-Oct;14(5):361-70. doi: 10.1177/036354658601400503. PMID 3535549
- [Background] Rayan F, Bhonsle S, Shukla DD. Clinical, MRI, and arthroscopic correlation in meniscal and anterior cruciate ligament injuries. Int Orthop. 2009 Feb;33(1):129-32. doi: 10.1007/s00264-008-0520-4. Epub 2008 Feb 23. PMID 18297284
- [Background] von Engelhardt LV, Lahner M, Klussmann A, Bouillon B, David A, Haage P, Lichtinger TK. Arthroscopy vs. MRI for a detailed assessment of cartilage disease in osteoarthritis: diagnostic value of MRI in clinical practice. BMC Musculoskelet Disord. 2010 Apr 20;11:75. doi: 10.1186/1471-2474-11-75. PMID 20406481